CLINICAL TRIAL: NCT00433576
Title: Phase I Repeat-Dose Study of Resveratrol in Colorectal Cancer Patients: Tolerability, Target Tissue Levels and Pharmacodynamics
Brief Title: Resveratrol in Treating Patients With Colorectal Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00864; NCI-2009-00864 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000528296; LRI-6930; N01-CN-25025; CCUM-TASK2B (Other: University of Michigan); N01-CN-25025-4 (Other: DCP); P30CA046592 (NIH)
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2011-10

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Stage I Colon Cancer; Stage I Rectal Cancer; Stage II Colon Cancer; Stage II Rectal Cancer; Stage III Colon Cancer; Stage III Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Resveratrol

ARMS (1):
- Treatment (resveratrol, colorectomy) (Experimental): STAGE I: Patients undergo an colorectal endoscopy. Patients whose biopsies confirm colorectal adenocarcinoma histology and require surgical resection continue on study stage 2.
  STAGE II: Patients receive oral resveratrol on days 1-8. Patients undergo colorectomy on day 9. A tumor biopsy is performed during endoscopy and colorectomy for research purposes.
  Interventions: Drug: resveratrol; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: resveratrol — Given orally
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of resveratrol in treating patients with colorectal cancer that can be removed by surgery. Resveratrol may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the relationship between oral dose of resveratrol and the colon mucosal levels of resveratrol and its metabolites in patients with resectable colorectal cancer.

II. Determine the relationship between colon mucosal levels of resveratrol and its metabolites and plasma concentrations of resveratrol and its metabolites in these patients.

III. Determine cyclooxygenase-2 (COX-2) expression in colorectal cancer tissue before and after treatment in these patients.

IV. Determine M_1G concentration in colonic cancer tissue and in circulating white blood cells (WBC) before and after treatment.

V. Correlate M_1G concentration in colorectal cancer tissue with M_1G concentration in circulating WBC.

VI. Assess the Ki67 labeling index in normal and malignant tissues in at least 10 fields per section.

VII. Correlate COX-2 expression in colorectal cancer tissue with COX-2 expression in circulating WBCs.

VIII. Assess the toxicity profile of this drug.

OUTLINE: This is a two-stage nonrandomized, open-label study. Patients are assigned to 1 of 2 dose levels in stage 2.

STAGE I: Patients undergo an colorectal endoscopy. Patients whose biopsies confirm colorectal adenocarcinoma histology and require surgical resection continue on study stage 2.

STAGE II: Patients receive oral resveratrol on days 1-8. Patients undergo colorectomy on day 9. A tumor biopsy is performed during endoscopy and colorectomy for research purposes.

Two biomarkers of the potential activity of resveratrol are measured in nonmalignant and malignant colorectal tissue biopsy samples: levels of M_1G adducts by immunoslot blot analysis and levels of cyclooxygenase-2 protein/Ki67 by immunohistochemistry. Blood samples are collected at baseline and during colorectomy for analysis of resveratrol and its metabolites and other pharmacokinetic studies.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1:

  * Radiological or clinical evidence of a colorectal malignancy
  * Requires colorectal endoscopy for diagnosis
* Stage 2:

  * Histologically confirmed adenocarcinoma of the colon or rectum by colorectal endoscopy in stage 1 study

    * Resectable disease
  * Planning to undergo colorectomy
* WHO performance status 0-2
* ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 1.5 mg/dL
* Hemoglobin ≥ 10 g/dL (transfusion allowed for anemia due to bleeding from the tumor)
* Suitable for general anesthesia
* No active peptic ulcer disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No excessive alcohol intake (more than UK recommended limit: 28 or 21 units per week for men or women, respectively)
* No other cancer that is currently under treatment, clinically detectable, or has been treated within the past 5 years (other than basal cell or squamous cell carcinomas)
* At least 6 months since prior and no concurrent participation in other invasive or drug studies
* No radiotherapy or chemotherapy within 4 weeks of endoscopic tissue sampling
* At least 24 hours since prior and no concurrent nonessential medications or nonsteroidal anti-inflammatory drugs
* No concurrent resveratrol-containing food and drink (e.g., wine, grapes, peanuts, mulberries, cranberries, blueberries, huckleberries)
* No concurrent vitamin supplements
* No concurrent chronic medications, including over-the-counter medications, that may interfere with the pharmacokinetics or pharmacodynamics measured
* No concurrent medication that could interfere with biomarker assay
* No concurrent anticoagulants including, warfarin and low molecular weight heparin
* No concurrent steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics of resveratrol | Up to 8 days
Concentrations of biomarkers | Up to day 9

CONTACTS AND LOCATIONS:
Overall Officials: Dean Brenner, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States